CLINICAL TRIAL: NCT06974214
Title: Patient- and Family-centred Care in the Adult Intensive Care Unit: a Feasibility Study
Acronym: FAM-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Søs Bohart, postdoc., Herlev Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Herlev Hospital
Record Dates: First submitted 2025-04-30; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Delirium; Anxiety; Post Intensive Care Unit Syndrome; Post Intensive Care Unit Syndrome Family; Depression; Posttraumatic Stress Disorder (PTSD); Mortality; Length of ICU Stay; Pain; Satisfaction Survey
Keywords: Patient- and family-centerede care; Feasibility; ICU
MeSH Terms: conditions — Delirium; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Pain

STUDY DESIGN:
Intervention Model Description: We will conduct a pre-/post two-group study design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual care (No Intervention): The group receives usual care.
- FAM-ICU intervention (Experimental): The group receives the FAM-ICU intervention
  Interventions: Other: FAM-ICU

INTERVENTIONS:
Other: FAM-ICU — This multi-component intervention comprises several concrete and manageable components and operationalizing patient- and family-centered care principles in clinical practice.
  Arms: FAM-ICU intervention

SUMMARY:
Background: In the intensive care unit (ICU), delirium in patients and long-term mental health challenges in both patients and their family members are highly prevalent. To address these issues, patient- and family-centered care has been recommended to alleviate the burdens associated with critical illness and ICU admission. We have developed the patient- and FAMily-centered care in the adult ICU intervention (FAM-ICU intervention). This multi-component intervention comprises several concrete and manageable components and operationalizing patient- and family-centered care principles in clinical practice. In this protocol, we describe a study aiming to evaluate the feasibility and acceptability of the FAM-ICU intervention in the adult ICU setting, including the feasibility of collecting relevant patient- and family-member outcome data.

Referenc: Bohart et al. 2024. Acta Anaesthesiol Scand

. 2025 Jan;69(1):e14539. doi: 10.1111/aas.14539. Epub 2024 Oct 24. Method: We will conduct a pre-/post two-group study design. We plan to recruit 30 adult ICU patients and their close family members at Herlev University Hospital in Denmark. The pre-group (n = 15) will receive usual care and the post-group (n = 15) will receive the FAM-ICU intervention. The FAM-ICU intervention involves interdisciplinary training of the ICU team and a systematic approach to information sharing and consultations with the patients and their family. Feasibility outcomes will include recruitment and retention rates, intervention fidelity, and the feasibility of participant outcome data collection. Acceptability will be assessed through questionnaires and interviews with clinicians, patients, and family members. Data collection is scheduled to begin in January 2025.

Discussion: This study will assess the feasibility and acceptability when implementing the FAM-ICU intervention and the feasibility of conducting a main trial to investigate its effectiveness on delirium in patients and the mental health of patients and family members. The data from the feasibility study will be used to guide sample size calculations, trial design, and final data collection methods for a subsequent stepped-wedge randomized controlled trial.

ELIGIBILITY:
Patients are eligible if they are:

* ≥18 years of age.
* Expected to require ICU admission for at least 48 hours in a mixed surgical and medical ICU for adult critically ill patients.

Family members are eligible if they are:

* ≥18 years of age.
* a close family member to a patient-enrolled in the FAM-ICU. A family-member can be blood-related or not. It may be a spouse, relative, partner, or friend as determined by the patient as a close family member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility, recruitment rate | during ICU admission.
  Number of approached participants who consent to participate.
Feasibility, Retention rate | 1 month post ICU admission
  The number of non-responders to the self-reported questionnaires at 6 months.
Feasibility, Fidelity | during ICU admission.
  The frequency and resource use of intervention delivery. Free text describing experienced barriers and facilitators for completing/not completing an intervention component.
Acceptability, Adherence | during ICU admission.
  Willingness to follow the intervention (Including barriers and facilitators).
Acceptability, Appropriateness | during ICU admission.
  Perception of how suitable the intervention is for the target population,
Acceptability, Convenience | during ICU admission.
  The intervention intrusiveness (how easy is it to apply)
Acceptability, effectiveness | during ICU admission.
  Perception of whether the intervention helps manage the problem.

SECONDARY OUTCOMES:
Free of delirium | during ICU admission.
  Number of delirium free days assessed by Confusion assessment method ICU (CAM-ICU)
Anxiety, patients | 1 month post ICU admission
  Symptoms of anxiety, using Hospital Anxiety and Depression Scale
Depression, patients | 1 month post ICU admission
  Symptoms of depression using Hospital Anxiety and Depression Scale.
PTSD, patients | 1 month post ICU admission
  Symptoms of PTSD using Harvard Trauma Questionnaire part 4 (HTQ-lV).
Health-related quality of life, patients | 1 month post ICU admission
  Assessed using EQ-5D
Free of life support | during ICU admission.
  Days without mechanical ventilation, receiving vasopressors and undergoing dialysis.
Survival | 1 month post ICU admission
  Days alive.
Employment status, patient | 1 month post ICU admission
  Employment as full-time, part-time, unemployed, self-employed, (paid/unpaid) on leave, student, or retired.
Cognitive function | 1 month post ICU admission
  Assessed using Mini Montreal Cognitive Assessment (Mini MoCA).
Out of hospital | 1 month post ICU admission
  Number of days out of hospital
Anxiety, family | 1 month post ICU admission
  Symptoms of anxiety using HADS
Depression, family | 1 post ICU admission
  Symptoms of depression using HADS
PTSD, family | 1 month post ICU admission
  Symptoms of PTSD using HTQ
Satisfaction, family | At ICU discharge.
  Survey for family-members regarding satisfaction.
Employment status, family | 1 month post ICU admission
  Employment as full-time, part-time, unemployed, self-employed, (paid/unpaid) on leave, student, or retired.
Anxiety, patients | 6 months post ICU
  Symptoms of anxiety, using Hospital Anxiety and Depression Scale
Depression, patients | 6 months post ICU
  Symptoms of depression using Hospital Anxiety and Depression Scale.
PTSD, patients | 6 months post ICU
  Symptoms of PTSD using Harvard Trauma Questionnaire part 4 (HTQ-lV).
Health-related quality of life, patients | 6 months post ICU
  Assessed using EQ-5D
Survival | 6 months post ICU
  Days alive.
Employment status, patient | 6 months post ICU
  Employment as full-time, part-time, unemployed, self-employed, (paid/unpaid) on leave, student, or retired.
Cognitive function | 6 months post ICU
  Assessed using Mini Montreal Cognitive Assessment (Mini MoCA).
Anxiety, family | 6 months post ICU
  Symptoms of anxiety using HADS
Depression, family | 6 months post ICU
  Symptoms of depression using HADS
PTSD, family | 6 months post ICU
  Symptoms of PTSD using HTQ
Employment status | 6 months post ICU
  Employment as full-time, part-time, unemployed, self-employed, (paid/unpaid) on leave, student, or retired.
Employment status, family | 6 months post ICU
  Employment as full-time, part-time, unemployed, self-employed, (paid/unpaid) on leave, student, or retired.
Out of hospital | 6 months post ICU
  Number of days out of hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bohart S, Waldau T, Andreasen AS, Moller AM, Thomsen T. Patient- and family-centered care in adult ICU (FAM-ICU): A protocol for a feasibility study. Acta Anaesthesiol Scand. 2025 Jan;69(1):e14539. doi: 10.1111/aas.14539. Epub 2024 Oct 24. PMID 39445615